CLINICAL TRIAL: NCT04003519
Title: Non-interventional, Prospective Study to Predict Lanreotide-induced Disease Activity Normalization in Acromegaly
Brief Title: Study to Predict Lanreotide-induced Disease Activity Normalization in Acromegaly
Acronym: PLAN-A
Status: Withdrawn | Type: Observational
Why Stopped: Study timeline delay, low site feasibility and delay concerns due to COVID-19.
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-DE-52030-368
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-06

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to collect data about predictive factors for the efficacy of Lanreotide Autogel in patients with acromegaly in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years and older with the capacity to consent
* Signed written informed consent
* Subject with hormonally active acromegaly defined by locally measured IGF-I levels 1.3 times above the age- and sex-adjusted normal range as determined at the last routine visit before baseline and after surgery
* Subject with the intention to be treated with lanreotide autogel according to the current local SmPC (Germany, Austria) prior to study enrolment

Exclusion Criteria:

* Participation in an interventional trial at the same time and/or within 3 months before baseline
* Subject represented by a legal guardian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects with biochemically active acromegaly, without previous treatment (medical treatment or radiotherapy) except for surgery and/or dopamine agonists (treatment terminated at or before baseline) who are already planned within the medical routine to be treated with lanreotide autogel.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-04 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with normalization of centrally assessed age and sex adjusted IGF-I levels at visit 4 (about 12 months) after treatment start with lanreotide autogel. | 12 months

SECONDARY OUTCOMES:
Proportion of subjects with normalization of centrally assessed age- and sex-adjusted IGF-I levels at visit 2, 3, and 5 after treatment start with lanreotide autogel | 3 , 6 and 18 months
Changes from baseline of centrally assessed IGF-I levels at visit 2, 3, 4, 5 after treatment start with lanreotide autogel | 3, 6, 12 and 18 months
Changes from baseline of centrally assessed random GH-levels at visit 2, 3, 4, 5 after treatment start with lanreotide autogel | 3, 6, 12 and 18 months
Changes from baseline of centrally assessed GH-BP levels at visit 2, 3, 4, 5 after treatment start with lanreotide autogel | 3, 6, 12 and 18 months
Proportion of subjects with GH-normalization - defined as centrally assessed random GH-levels (GH < 1 μg/L) - at visits 2, 3, 4, and 5 during treatment with lanreotide autogel. | 3, 6, 12 and 18 months
Predictors for reduction of age- and sex-adjusted IGF-I to normal levels (control of acromegaly) at visits 4 compared to baseline and Last Visit Available (LVA) compared to baseline. | baseline and 12 months
Predictors of change in IGF-I between baseline compared to visit 4 and baseline compared to LVA. | baseline and 12 months
Predictors of change in random GH-levels between baseline compared to visit 4 and baseline compared to LVA | baseline and 12 months
Patient's global impression of change (PGIC) | 3, 6, 12 and 18 months
  Scale is used to assess the validity of Patient Global Impression of Change (PGIC). the score ranges between 1= very much worse and 7 = very much improved
Changes in signs and symptoms (Numerical Rating Scale), patient's global impression of change (PGIC) | Baseline, 3, 6, 12 and 18 months
  It will be measured using Numerical Rating Scale to assess the average presence or severity of the symptoms. The score ranges from 0 = no symptom at all to 10 = maximum intensity of the symptom
Quality of life between baseline and visits 2, 3, 4 and 5. | Baseline, 3, 6, 12 and 18 months
  Measured by a generic, multipurpose short-form survey with 12 questions (SF-12). Scale provides information about mental and physical functioning and overall health-related-QoL. ". Higher scores indicate a better QoL.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen